CLINICAL TRIAL: NCT03898596
Title: Umbilical Vessel Catheterization Under ECG Monitoring and Guidance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 49778
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pediatric ALL
Keywords: Neonates; Electrocardiogram; Umbilical Vein Catheterization
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ECG Monitoring (Other): ECG readings will be collected for neonatal patients who require or currently have UVC
  Interventions: Diagnostic Test: ECG

INTERVENTIONS:
Diagnostic Test: ECG — An ECG collects superficial readings of heart activity

SUMMARY:
Umbilical venous catheters (UVC) are typically places with poor guidance and some radiological confirmation. Misplacement of the catheter could lead to its placement in other unintended anatomical areas such as the liver or the spleen, which could be detrimental in critically-ill infants. Our study aims at using a more non-invasive means of placing and continuously monitoring catheter placement using superficial electrocardiogram (ECG) tracings.

ELIGIBILITY:
Inclusion Criteria:

* Neonate pediatric patient
* 2 - 6kg
* Require or currently have UVC

Exclusion Criteria:

* Participants who do not consent or have parental consent
* Patients who are clinically unstable

Ages: 1 Day to 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram Readings | Duration of ECG placement and reading (typically 15 minutes)
  A normal heart rhythm contains a P wave, a QRS, and a T wave. Readings will include amplitude, deflection, and duration of such elements to record electrical heart activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No